CLINICAL TRIAL: NCT06401291
Title: The Novel Use of Transcutaneous Electrical Nerve Stimulation in Patients With Angina and Non-Obstructive Coronary Arteries: a Pilot Study
Brief Title: Transcutaneous Electrical Nerve Stimulation in Patients With Angina and Non-Obstructive Coronary Arteries
Acronym: TENS-ANOCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Inge Wijnbergen, MD, PhD, Catharina Ziekenhuis Eindhoven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL84910.100.23
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Microvascular Angina; Vasospastic Angina
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris, Variant | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: All patients who meet the inclusion criteria will receive TENS treatment for a period of 1 month. At baseline and at 1 month evaluation will take place.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label (Other): See intervention: all patients included in the study will receive TENS treatment for a period of 1 month
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — Device consists of two electrodes that are applied to the chest region and are connected to a battery operated TENS (Frequency 80Hz, pulse width 150us and amplitude variable (patient dependent)). The device will be used a minimum of three times daily for 30 minutes and additionally during symptoms.
  Other Names: TENS

SUMMARY:
In patients with angina pectoris undergoing a coronary angiography (CAG) up to 40% do not have obstructive coronary artery disease (CAD). The majority of patients with no obstructive CAD are women with a frequency of up to 70% compared to 50% in men. These patients are diagnosed as having angina and non-obstructive coronary arteries (ANOCA). There are two endotypes of ANOCA. The first endotype is microvascular angina (MVA) caused by a combination of structural microcirculatory remodelling and functional arteriolar dysregulation, also called coronary microvascular dysfunction (CMD). The second endotype is vasospastic angina (VSA) caused by epicardial coronary artery spasm that occurs when a hyper-reactive epicardial coronary segment is exposed to a vasoconstrictor stimulus. Both endotypes of ANOCA are associated with significantly greater one-year risk of myocardial infarction (MI) and all-cause mortality, have a significantly impaired quality of life and have a high health care resource utilisation.

The current treatment for ANOCA consists of three aspects. The first aspect is managing lifestyle factors such as weight management, smoking cessation and exercise. The second aspect is managing known cardiovascular risk factors such as hypertension, dyslipidaemia and diabetes mellitus. And the third aspect is antianginal medication. In both endotypes ACE inhibitors or angiotensin II receptor blockers should be considered. In MVA the antianginal medication that can be used are betablocker, calcium channel blocker, nicorandil, ranolazine, ivabradine and/or trimetazidine. In VSA calcium channel blocker, long-acting nitrate and/or nicorandil can be initiated as antianginal therapy. Despite these treatment option approximately 25% of ANOCA patients have refractory angina symptoms.

A possible treatment modality for ANOCA patients with refractory angina pectoris is spinal cord stimulation (SCS) or transcutaneous electrical nerve stimulation (TENS). Previous research (in patients with cardiac syndrome X) has shown that SCS improves time until angina and ischaemia, significantly less angina and an improvement in quality of life. These findings suggest that SCS and/or TENS could be a possible treatment modality for patients with ANOCA.

The aim of this pilot study is to investigate whether treatment with TENS during a one month period leads to a significant reduction of angina pectoris and therefore a significant improvement in quality of life in patients with proven ANOCA, encompassing both endotypes (MVA and VSA).

ELIGIBILITY:
Inclusion Criteria:

* Angina and no obstructive coronary artery disease (ANOCA) (CCS class III or IV)
* Microvascular angina (MVA):

  * FFR > 0.8
  * CFR < 2.0
  * IMR ≥ 25
* Vasospastic angina (VSA):

  * FFR > 0.8
  * CFR ≥ 2.0
  * IMR < 25
  * During acetylcholine testing: ≥ 90% diameter reduction, angina pectoris and ischaemic ECG changes
* Persisting angina pectoris despite optimal medical therapy (OMT) defined as:

  * MVA: Betablocker, calcium channel blocker, nicorandil and/or ivabradine (Important side note: ranolazine and trimetazidine cannot be prescribed in the Netherlands).
  * VSA: Calcium channel blocker, long-acting nitrate and/or nicorandil. In the maximum tolerated dose. If the patient is currently not using one of the medications due to side-effects, this should be clearly stated.
* Age > 18 years

Exclusion Criteria:

* Both endotypes (VSA and MVA) present based on CFT findings.
* Inability to give informed consent
* Inability to perform a 6-minute walking test
* The presence of a cardiac implanted electronic device (CIED); pacemaker and/or Implantable Cardiac Defibrillator (ICD). Due to the risk of interference between TENS and CIED
* Presence of a spinal cord stimulator for another indication such as complex regional pain syndrome, failed back surgery syndrome, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in summary score of Seattle Angina Questionnaire | Baseline; 1 month
  Change in the summary score of the Seattle Angina Questionnaire (SS SAQ) after 1 month treatment with TENS, compared to baseline.

SECONDARY OUTCOMES:
Change in physical limitations domain of Seattle Angina Questionnaire | Baseline; 1 month
  Change in physical limitations domain of the Seattle Angina Questionnaire (PL SAQ) after 1 month treatment with TENS, compared to baseline.
Change in angina frequency domain of Seattle Angina Questionnaire | Baseline; 1 month
  Change in angina frequency domain of the Seattle Angina Questionnaire (AF SAQ) after 1 month treatment with TENS, compared to baseline.
Change in angina stability domain of Seattle Angina Questionnaire | Baseline; 1 month
  Change in angina stability domain of the Seattle Angina Questionnaire (AS SAQ) after 1 month treatment with TENS, compared to baseline.
Change in treatment satisfaction domain of Seattle Angina Questionnaire | Baseline; 1 month
  Change in treatment satisfaction domain of the Seattle Angina Questionnaire (TS SAQ) after 1 month treatment with TENS, compared to baseline.
Change in quality of life domain of Seattle Angina Questionnaire | Baseline; 1 month
  Change in quality of life domain of the Seattle Angina Questionnaire (QoL SAQ) after 1 month treatment with TENS, compared to baseline.
Changes in patient condition | Baseline; 1 month
  Change in patient condition using the 6-minute walking test after 1 month treatment with TENS, compared to baseline
Change in CCS class | Baseline; 1 month
  Change in grading of angina pectoris using the Canadian Cardiovascular Society (CCS) class after 1 month treatment with TENS compared to baseline

OTHER OUTCOMES:
Side effects of TENS use | 1 month
  Register all side effects (such as skin irritation, tenderness and/or TENS discomfort) experienced by the patient over the 1 month treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No